CLINICAL TRIAL: NCT02679742
Title: The PSSMAR Study (Postacute Sarcopenia, Supplementation With β-hydroxyMethylbutyrate After Resistance Training)
Brief Title: Postacute Sarcopenia: Supplementation With β-hydroxyMethylbutyrate After Resistance Training
Acronym: PSSMAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSSMAR 2015/6288/I
Record Dates: First submitted 2016-01-26; First posted 2016-02-10 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2020-04

CONDITIONS: Sarcopenia
Keywords: beta hydroxy beta methylbutyrate; older people; muscle mass; muscle strength; post-acute
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- β-hydroxymethylbutyrate (Experimental): β-hydroxymethylbutyrate 3 grams once a day combined with a resistance training program
  Interventions: Dietary Supplement: β-hydroxymethylbutyrate
- Placebo (Placebo Comparator): Maltodextrin 3 grams once a day combined with a resistance training program
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: β-hydroxymethylbutyrate — β-hydroxymethylbutyrate 3 grams once a day combined with a resistance training program (3 progressive resistance training sessions per week) during 12 weeks
  Arms: β-hydroxymethylbutyrate
Dietary Supplement: Placebo — Maltodextrin 3 grams once a day combined with a resistance training program (3 progressive resistance training sessions per week) during 12 weeks
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled, parallel study to assess the effects of β-hydroxymethylbutyrate (β-HMB) combined with a resistance training program, after an acute process in older patients with sarcopenia in terms of muscle mass, muscle strength and physical performance. Treatments compared will be β-hydroxymethylbutyrate (β-HMB) with a resistance training program or placebo with a resistance training program.

DETAILED DESCRIPTION:
Sarcopenia is a geriatric syndrome characterized by the loss of skeletal muscle mass and strength that occurs with advancing age; it is related to frailty, falls, worsening quality of life, and death in chronic and elderly patients. Diagnosis of sarcopenia is based on clinical criteria: presence of low muscle mass and the presence of low muscle function and/or low physical performance. The latest developments indicate that dietary supplementation combined with resistance exercise could be an option to improve muscle mass and function.

The objective of the study is to assess the effects of β-hydroxymethylbutyrate (β-HMB) combined with a resistance training program, after an acute process in older patients with sarcopenia in terms of muscle mass, muscle strength and physical performance.

Design: A randomized, double-blind, placebo-controlled, parallel study with two intervention groups. The investigators shall compare placebo against an intervention with β-HMB in patients performing a resistance training program after an acute process (post-acute period) during 12 weeks. There will be 16 patients in each arm of the study. Additionally a one year follow up visit will be performed.

ELIGIBILITY:
Inclusion Criteria:

* male or female ≥60 years old
* sarcopenia diagnosis and case-finding criteria following European Working Group On Sarcopenia in Older People (EWGSOP)
* being discharged from post-acute care geriatric unit for rehabilitation treatment
* ambulatory prior to the recent acute process
* cognitive situation that let them to understand and follow an active physical rehabilitation program (Mini-Mental Status Examination ≥21/30)
* voluntary participation and being able and willing to provide an informed consent

Exclusion Criteria:

* potential participants will be excluded if they have active malignancy (exception basal or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix)
* major lower limb surgery over the past 6 months (knee or hip arthroplasty)
* contraindication for resistance training
* performed regular exercise in the last 6 months
* use of any medications interfering with the nutritional intervention
* serious clinical conditions that compromises and endanger the patient's life
* contraindication, intolerance or allergy to β-hydroxymethylbutyrate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline handgrip strength at 12 weeks | From baseline till 12 weeks
  Handgrip strength will be measured by a hand-held dynamometer (JAMAR®, Nottinghamshire, UK) and expressed in Kg
Change from baseline physical performance-gait speed- at 12 weeks | From baseline till 12 weeks
  Physical performance will be assessed with gait speed in the 4-m walk test
Change from baseline physical performance-SPPB- at 12 weeks | From baseline till 12 weeks
  Physical performance will be assessed with gait speed in short physical performance battery

SECONDARY OUTCOMES:
Number of hospital readmissions | From baseline till 12 weeks
  Admissions in acute care due to medical health issues
Change from baseline functional status at 12 weeks | From baseline till 12 weeks
  Functional status assessed by the Barthel index
Absolute functional gain in 12 weeks | From baseline till 12 weeks
  Absolute functional gain measured with Barthel scale
Relative functional gain in 12 weeks | From baseline till 12 weeks
  Relative functional gain measured with Barthel scale
Change from baseline rehabilitation impact indices at 12 weeks | From baseline till 12 weeks
  Rehabilitation Efficiency Index
Number of adverse events | From baseline till 12 weeks
  Adverse events will be collected by medical interview during the study
Change from baseline lean and fat body mass (muscle mass) at 12 weeks | From baseline till 12 weeks
  Lean and fat body mass will be measured by electrical impedance measured in kg and expressed as normal, low or high values according to normality values for the European population

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dolores Sánchez-Rodríguez, PhD, MD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital de l'Esperanza, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Rodriguez D, Marco E, Ronquillo-Moreno N, Miralles R, Mojal S, Vazquez-Ibar O, Escalada F, Muniesa JM. The PSSMAR study. Postacute sarcopenia: Supplementation with beta-hydroxyMethylbutyrate after resistance training: Study protocol of a randomized, double-blind controlled trial. Maturitas. 2016 Dec;94:117-124. doi: 10.1016/j.maturitas.2016.08.019. Epub 2016 Sep 9. No abstract available. PMID 27823730
- [Background] Reginster JY, Beaudart C, Al-Daghri N, Avouac B, Bauer J, Bere N, Bruyere O, Cerreta F, Cesari M, Rosa MM, Cooper C, Cruz Jentoft AJ, Dennison E, Geerinck A, Gielen E, Landi F, Laslop A, Maggi S, Prieto Yerro MC, Rizzoli R, Sundseth H, Sieber C, Trombetti A, Vellas B, Veronese N, Visser M, Vlaskovska M, Fielding RA. Update on the ESCEO recommendation for the conduct of clinical trials for drugs aiming at the treatment of sarcopenia in older adults. Aging Clin Exp Res. 2021 Jan;33(1):3-17. doi: 10.1007/s40520-020-01663-4. Epub 2020 Jul 31. PMID 32737844
- [Background] Sanchez-Rodriguez D, Marco E, Miralles R, Guillen-Sola A, Vazquez-Ibar O, Escalada F, Muniesa JM. Does gait speed contribute to sarcopenia case-finding in a postacute rehabilitation setting? Arch Gerontol Geriatr. 2015 Sep-Oct;61(2):176-81. doi: 10.1016/j.archger.2015.05.008. Epub 2015 May 29. PMID 26051706
- [Background] Sanchez-Rodriguez D, Marco E, Miralles R, Fayos M, Mojal S, Alvarado M, Vazquez-Ibar O, Escalada F, Muniesa JM. Sarcopenia, physical rehabilitation and functional outcomes of patients in a subacute geriatric care unit. Arch Gerontol Geriatr. 2014 Jul-Aug;59(1):39-43. doi: 10.1016/j.archger.2014.02.009. Epub 2014 Mar 1. PMID 24726179
- [Background] Sanchez-Rodriguez D, Marco E, Cruz-Jentoft AJ. Defining sarcopenia: some caveats and challenges. Curr Opin Clin Nutr Metab Care. 2020 Mar;23(2):127-132. doi: 10.1097/MCO.0000000000000621. PMID 31789867
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Sanchez-Rodriguez D, Marco E, Davalos-Yerovi V, Lopez-Escobar J, Messaggi-Sartor M, Barrera C, Ronquillo-Moreno N, Vazquez-Ibar O, Calle A, Inzitari M, Piotrowicz K, Duran X, Escalada F, Muniesa JM, Duarte E. Translation and Validation of the Spanish Version of the SARC-F Questionnaire to Assess Sarcopenia in Older People. J Nutr Health Aging. 2019;23(6):518-524. doi: 10.1007/s12603-019-1204-z. PMID 31233072
- [Derived] Meza-Valderrama D, Sanchez-Rodriguez D, Messaggi-Sartor M, Munoz-Redondo E, Morgado-Perez A, Tejero-Sanchez M, De Jaime-Gil E, Leiva-Banuelos N, Marco E. Supplementation with beta-hydroxy-beta-methylbutyrate after resistance training in post-acute care patients with sarcopenia: A randomized, double-blind placebo-controlled trial. Arch Gerontol Geriatr. 2024 Apr;119:105323. doi: 10.1016/j.archger.2023.105323. Epub 2023 Dec 27. PMID 38171034